CLINICAL TRIAL: NCT06624228
Title: A Multicenter, Randomized, Double-Blind, Risankizumab-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Study Participants With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Study Participants With Active Psoriatic Arthritis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA0016; 2024-511738-11 (Registry Identifier: EU Clinical Trials); U1111-1306-6697 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis
Keywords: bimekizumab; risankizumab; arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis | interventions — bimekizumab; risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bimekizumab (Experimental): Study participants will receive assigned bimekizumab dosage regimen and placebo to maintain the blinding during treatment period.
  Interventions: Drug: Bimekizumab; Drug: Placebo
- Risankizumab (Active Comparator): Study participants will receive assigned risankizumab dosage regimen and placebo to maintain the blinding during treatment period.
  Interventions: Drug: Risankizumab; Drug: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Study participants will receive bimekizumab at pre-specified time points.
  Arms: Bimekizumab
Drug: Risankizumab — Study participants will receive risankizumab at pre-specified time points.
  Arms: Risankizumab
Drug: Placebo — Study participants will receive placebo at pre-specified time points.

SUMMARY:
The purpose of the study is to compare the efficacy of bimekizumab versus risankizumab after 16 weeks of treatment in study participants with active psoriatic arthritis (PsA).

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have a documented diagnosis of adult-onset PsA classified by and that meets the CASPAR classification criteria for at least 6 months prior to Screening with active PsA (despite previous csDMARD or apremilast therapy) and must have at Baseline tender joint count (TJC) ≥3 out of 68 joints and swollen joint count (SJC) ≥3 out of 66 joints (dactylitis of a digit counts as 1 joint each).
* Study participant must have at least 1 active psoriatic lesion(s) and/or a documented history of chronic plaque-type psoriasis (PSO).
* Study participants may currently be on conventional synthetic disease-modifying antirheumatic drug (csDMARD) therapy and must have previously been treated with at least 1 csDMARD (methotrexate (MTX), leflunomide (LEF), sulfasalazine (SSZ)). Study participants must have had an inadequate response to therapy or discontinued due to intolerance. (Inadequate response is determined by the Investigator and is defined as not achieving the minimal response after 12 weeks of therapy.)
* Study participants can either be biological disease-modifying antirheumatic drug (bDMARD)-naïve or have received not more than 1 prior tumor necrosis factor alpha (TNFα) inhibitor. Study participants who have been on a TNFα inhibitor previously must not have discontinued the TNFα inhibitor due to financial or health insurance reasons and must have either:
* experienced an inadequate response to previous treatment given at an approved dose for at least 3 months, or
* been intolerant to administration (eg, had a side-effect/adverse event (AE) that led to discontinuation).

Exclusion Criteria:

* Study participant has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the study participant's ability to participate in this study.
* Female participants who are breastfeeding, pregnant, or plan to become pregnant during the study.
* Participant has an active infection or a history of recent serious infections.
* Participant has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection.
* Study participant has a diagnosis of inflammatory conditions other than PSO or PsA including, but not limited to, rheumatoid arthritis, sarcoidosis, systemic lupus erythematosus, reactive arthritis, and axial spondyloarthritis.
* Study participants with a history of anterior uveitis are allowed if they have no active symptoms at Screening or Baseline. Study participants with a diagnosis of Crohn's disease or ulcerative colitis are allowed if they have no active symptomatic disease at Screening or Baseline.
* Study participants with fibromyalgia or osteoarthritis symptoms that in the Investigator's opinion would have potential to interfere with efficacy assessments.
* Participant has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer.
* Participant has a history of chronic alcohol or drug abuse within 6 months prior to Screening.
* Study participants taking psoriatic arthritis (PsA) medications other than MTX, SSZ, apremilast, hydroxychloroquine (HCQ), LEF, nonsteroidal anti-inflammatory drug (NSAIDs)/ cyclooxygenase-2 (COX-2) inhibitors, oral corticosteroids, and analgesics as outlined in the Inclusion criteria.
* Study participant is taking or has taken prohibited PsA or PSO medications without meeting the mandatory wash-out period relative to the Baseline Visit.
* Study participant is taking or has taken janus kinase (JAK) inhibitor.
* Study participant is taking or has taken bDMARDs, including bimekizumab or risankizumab, with the exception of having received 1 prior TNFα inhibitor.
* Study participant previously participated in another study of a medical device under investigation within the 4 weeks prior to the Screening Visit or is currently participating in another study of a medical device under investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-05-26 (Estimated)

PRIMARY OUTCOMES:
American College of Rheumatology 50 (ACR50) at Week 16 | Week 16
  The ACR50 response rate is based on a 50% or greater improvement of arthritis relative to Baseline.
  * TJC and SJC: 2-point scale (0=absent;1=present) • Patient's Global Assessment of Psoriatic Arthritis (PGA-PsA): 100 VAS (0=very good, no symptoms;100=very poor, severe symptoms)
  * Physician's Global Assessment of Psoriatic Arthritis (PhGA-PsA): 100 VAS (0=very good, asymptomatic, no limitation of normal activities;100=very poor, very severe symptoms which were intolerable, inability to carry out all normal activities). • Patient's Assessment of Arthritis Pain (PtAAP): 100 VAS (0=no pain;100=most severe pain).
  * Health Assessment Questionnaire Disability Index score (HAQ-DI) assessed degree of difficulty experienced in 8 domains of daily living activities (20 questions), total score (0-3) computed from item scores, with lower scores meaning less disability.
  * High sensitivity C-reactive protein (hs-CRP) in mg/L

SECONDARY OUTCOMES:
Minimal Disease Activity (MDA) at Week 16 | Week 16
  A study participant is considered as having MDA if 5 or more of the following 7 criteria are fulfilled:
  * Tender joint count ≤1
  * Swollen joint count ≤1
  * PASI ≤1 or BSA ≤3
  * PtAAP VAS ≤15
  * PGA-PsA VAS ≤20
  * HAQ-DI ≤0.5
  * Tender enthesial points ≤1
Percentage of participants reaching the composite endpoint composed of ACR50 and Psoriasis Area and Severity Index 100% (PASI100) response at Week 16 in the subgroup of study participants with PSO involving at least 3% body surface area (BSA) at Baseline | Week 16
  The ACR50 response rate is based on a 50% or greater improvement of arthritis relative to Baseline.
  The PASI100 response is based on at least 100% improvement in the PASI score. Body divided into 4 areas: head, upper extremities, trunk and lower extremities. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Incidence of Participants With Treatment-emergent adverse events (TEAEs) | From Baseline (Day 1) to End of Safety Follow-Up (up to 42 weeks)
  An Adverse Event (AE) is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of investigational medicinal product (IMP), whether or not considered related to the IMP.
Incidence of Participants With Treatment-emergent serious AEs | From Baseline (Day 1) to End of Safety Follow-Up (up to 42 weeks)
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization Is a congenital anomaly or birth defect
  * Results in permanent or significant disability/incapacity
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Incidence of Participants With TEAEs leading to withdrawal from investigational medicinal product (IMP) | From Baseline (Day 1) to End of Safety Follow-Up (up to 42 weeks)
  An AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of IMP, whether or not considered related to the IMP.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (127):
- United States (34):
  - Pa0016 50662, Gilbert, Arizona
  - Pa0016 50062, Glendale, Arizona
  - Pa0016 50058, Phoenix, Arizona
  - Pa0016 50131, Sun City, Arizona
  - Pa0016 50654, Covina, California
  - Pa0016 50663, San Diego, California
  - Pa0016 50672, Santa Monica, California
  - Pa0016 50630, Clearwater, Florida
  - Pa0016 50679, Cutler Bay, Florida
  - Pa0016 50685, Fort Lauderdale, Florida
  - Pa0016 50059, Ormond Beach, Florida
  - Pa0016 50324, Plantation, Florida
  - Pa0016 50678, Zephyrhills, Florida
  - Pa0016 50651, Skokie, Illinois
  - Pa0016 50650, Willowbrook, Illinois
  - Pa0016 50686, Hagerstown, Maryland
  - Pa0016 50665, Lansing, Michigan
  - Pa0016 50551, Saint Clair Shores, Michigan
  - Pa0016 50689, Eagan, Minnesota
  - Pa0016 50682, Kansas City, Missouri
  - Pa0016 50016, St Louis, Missouri
  - Pa0016 50653, Albuquerque, New Mexico
  - Pa0016 50666, Brooklyn, New York
  - Pa0016 50664, Middletown, Ohio
  - Pa0016 50680, Vandalia, Ohio
  - Pa0016 50652, Duncansville, Pennsylvania
  - Pa0016 50006, Wyomissing, Pennsylvania
  - Pa0016 50001, Jackson, Tennessee
  - Pa0016 50673, Fort Worth, Texas
  - Pa0016 50048, Katy, Texas
  - Pa0016 50657, Lubbock, Texas
  - Pa0016 50655, Tomball, Texas
  - Pa0016 50061, Spokane Valley, Washington
  - Pa0016 50674, Glendale, Wisconsin
- Australia (6):
  - Pa0016 30002, Clayton
  - Pa0016 30034, Footscray
  - Pa0016 30033, Heidelberg
  - Pa0016 30003, Maroochydore
  - Pa0016 30032, Parramatta
  - Pa0016 30009, Westmead
- Bulgaria (11):
  - Pa0016 40313, Pleven
  - Pa0016 40006, Plovdiv
  - Pa0016 40813, Plovdiv
  - Pa0016 40818, Plovdiv
  - Pa0016 40820, Plovdiv
  - Pa0016 40656, Rousse
  - Pa0016 40823, Rousse
  - Pa0016 40314, Sofia
  - Pa0016 40380, Sofia
  - Pa0016 40811, Sofia
  - Pa0016 40819, Sofia
- Canada (2):
  - Pa0016 50041, Québec
  - Pa0016 50044, Trois-Rivières
- Czechia (7):
  - Pa0016 40065, Brno
  - Pa0016 40062, Moravska Ostrava A Privoz
  - Pa0016 40802, Ostrava
  - Pa0016 40066, Prague
  - Pa0016 40801, Prague
  - Pa0016 40010, Uherské Hradiště
  - Pa0016 40012, Zlín
- Germany (9):
  - Pa0016 40073, Bad Nauheim
  - Pa0016 40025, Berlin
  - Pa0016 40138, Bonn
  - Pa0016 40808, Cologne
  - Pa0016 40072, Freiburg im Breisgau
  - Pa0016 40029, Hamburg
  - Pa0016 40810, Herne
  - Pa0016 40724, München
  - Pa0016 40800, Ratingen
- Hungary (4):
  - Pa0016 40081, Budapest
  - Pa0016 40804, Budapest
  - Pa0016 40809, Hódmezővásárhely
  - Pa0016 40031, Szeged
- Japan (9):
  - Pa0016 20035, Bunkyō City
  - Pa0016 20043, Itabashi-ku
  - Pa0016 20045, Kita-gun
  - Pa0016 20049, Kitakyushu
  - Pa0016 20069, Meguro-ku
  - Pa0016 20336, Mitaka-shi
  - Pa0016 20041, Osaka
  - Pa0016 20046, Osaka
  - Pa0016 20031, Sapporo
- Poland (30):
  - Pa0016 40789, Bialystok
  - Pa0016 40791, Bialystok
  - Pa0016 40824, Bialystok
  - Pa0016 40119, Bydgoszcz
  - Pa0016 40798, Bydgoszcz
  - Pa0016 40038, Elblag
  - Pa0016 40795, Katowice
  - Pa0016 40092, Krakow
  - Pa0016 40490, Krakow
  - Pa0016 40502, Krakow
  - Pa0016 40792, Krakow
  - Pa0016 40037, Lublin
  - Pa0016 40483, Nadarzyn
  - Pa0016 40091, Nowa Sól
  - Pa0016 40796, Olsztyn
  - Pa0016 40794, Opole
  - Pa0016 40044, Poznan
  - Pa0016 40090, Poznan
  - Pa0016 40807, Poznan
  - Pa0016 40790, Sochaczew
  - Pa0016 40788, Torun
  - Pa0016 40094, Warsaw
  - Pa0016 40394, Warsaw
  - Pa0016 40539, Warsaw
  - Pa0016 40604, Warsaw
  - Pa0016 40793, Warsaw
  - Pa0016 40797, Warsaw
  - Pa0016 40043, Wroclaw
  - Pa0016 40095, Wroclaw
  - Pa0016 40805, Wroclaw
- Spain (8):
  - Pa0016 40806, A Coruña
  - Pa0016 40269, Bilbao
  - Pa0016 40231, Madrid
  - Pa0016 40102, Málaga
  - Pa0016 40803, Sabadell
  - Pa0016 40753, Santiago de Compostela
  - Pa0016 40049, Seville
  - Pa0016 40799, Seville
- United Kingdom (7):
  - Pa0016 40833, Barnet
  - Pa0016 40281, Leeds
  - Pa0016 40827, Luton
  - Pa0016 40237, Manchester
  - Pa0016 40306, Newcastle upon Tyne
  - Pa0016 40828, Reading
  - Pa0016 40108, Salford

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed.All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org